CLINICAL TRIAL: NCT06128551
Title: Phase 1b/2, Multicenter, Open-label, Dose Escalation and Dose Expansion Study of Elironrasib and Daraxonrasib as Monotherapies and Combination Therapy in Patients With Advanced KRAS G12C-Mutated Solid Tumors
Brief Title: Study of Elironrasib and Daraxonrasib as Monotherapies and Combination Therapy in Participants With Advanced KRAS G12C Mutant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RMC-6291-101
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Colorectal Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: RMC-6291; RAS (ON); KRAS; KRASG12C; KRASG12C (ON); Targeted therapy; Metastatic Cancer; Lung Cancer; Lung Neoplasms; Thoracic Neoplasms; Non-small Cell Lung Cancer; Carcinoma, Non-Small Cell Lung; NSCLC; Colorectal Cancer; Colonic Neoplasms; CRC; Appendiceal Cancer; KRAS mutation; STK11/LKB1; KEAP1; Bronchial neoplasms; Respiratory tract neoplasms; Neoplasms by site; Neoplasms; Colon Cancer; Rectal Cancer; Lung disease; Respiratory tract diseases; Pancreatic Cancer; Carcinoma, Pancreatic Ductal; PDAC; Gastrointestinal Neoplasms; Intestinal Neoplasms; Esophageal Cancer; Ampullary Cancer; Gastric Cancer; Gynecological Cancer; Ovarian Cancer; Endometrial Cancer; RMC-6236; Elironrasib; Daraxonrasib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasm Metastasis; Lung Neoplasms; Thoracic Neoplasms; Colonic Neoplasms; Appendiceal Neoplasms; Bronchial Neoplasms; Respiratory Tract Neoplasms; Neoplasms by Site; Neoplasms; Rectal Neoplasms; Lung Diseases; Respiratory Tract Diseases; Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal; Gastrointestinal Neoplasms; Intestinal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Elironrasib Monotherapy (Experimental): Phase 2 only
  Interventions: Drug: Elironrasib
- Daraxonrasib Monotherapy (Experimental): Phase 2 only
  Interventions: Drug: Daraxonrasib
- Daraxonrasib + Elironrasib Combination (Experimental): Phase 1b and 2
  Interventions: Drug: Elironrasib; Drug: Daraxonrasib

INTERVENTIONS:
Drug: Elironrasib — oral tablets
  Other Names: RMC-6291
  Arms: Daraxonrasib + Elironrasib Combination; Elironrasib Monotherapy
Drug: Daraxonrasib — oral tablets
  Other Names: RMC-6236
  Arms: Daraxonrasib + Elironrasib Combination; Daraxonrasib Monotherapy

SUMMARY:
This study is to evaluate the safety, tolerability, and PK profiles of Elironrasib and Daraxonrasib as monotherapies and combination therapy in patients with KRAS G12C-mutated solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1b/2 study evaluating elironrasib and daraxonrasib, administered as monotherapy and in combination, in patients with advanced KRAS G12C-mutated solid tumors to determine the maximum tolerated dose (MTD), identify the recommended Phase 2 dose and schedule (RP2DS), and preliminarily assess antitumor activity.

The study includes a Phase 1b dose escalation and expansion of combination therapy, followed by a Phase 2 evaluation of the selected RP2DS as monotherapy and combination therapy to further assess safety and antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Histology: pathologically documented, KRAS G12C-mutated, advanced or metastatic solid tumors not amendable to curative therapy

  1. Phase 1b Dose Escalation: solid tumors, previously treated
  2. Phase 1b Dose Expansion and Phase 2:

  i. NSCLC, previously treated with immunotherapy, chemotherapy, and KRAS G12C (OFF) inhibitors ii. Solid tumors, previously treated, naïve to KRAS G12C (OFF) inhibitors.
* ECOG performance status 0 or 1
* Adequate organ function

Exclusion Criteria:

* Primary central nervous system (CNS) tumors
* Active brain metastases
* Known impairment of GI function that would alter the absorption
* Major surgical procedures within 28 days or non-study related minor procedures within 7 days of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) in Phase 1b | Up to approximately 3 years
  Incidence and severity of treatment-emergent AEs and serious AEs as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5
Changes in vital signs in Phase 1b | Up to approximately 3 years
  Number of patients with clinically significant changes in vital signs
Changes in clinical laboratory test values in Phase 1b | Up to approximately 3 years
  Number of patients with clinically significant changes in clinical laboratory test values
Dose Limiting Toxicities in Phase 1b | 21 days
  Number of participants with dose limiting toxicities
Changes in ECGs in Phase 1b | Up to approximately 3 years
  Number of patients with clinically significant changes in ECGs
Overall Response Rate (ORR) in Phase 2 | Up to approximately 3 years
  Overall response rate per RECIST v1.1 as assessed by blinded independent central review (BICR)

SECONDARY OUTCOMES:
Maximum Observed Blood Concentration of Elironrasib and Daraxonrasib | up to 21 weeks
  Cmax
Time to Reach Maximum Blood Concentration of Elironrasib and Daraxonrasib | up to 21 weeks
  Tmax
Area Under Blood Concentration Time Curve of Elironrasib and Daraxonrasib | up to 21 weeks
  AUC
Elimination Half-Life of Elironrasib and Daraxonrasib | up to 21 weeks
  t1/2
Ratio of accumulation of Elironrasib and Daraxonrasib from a single dose to steady state with repeated dosing | up to 21 weeks
  accumulation ratio
Overall Response Rate (ORR) in Phase 1b | Up to approximately 3 years
  Overall response rate per RECIST v1.1
Duration of Response (DOR) | Up to approximately 3 years
  Duration of response per RECIST v1.1
Disease Control Rate in Phase 1b | Up to approximately 3 years
  Disease Control rate per RECIST v1.1
Time to Response (TTR) in Phase 1b | Up to approximately 3 years
  Time to response per RECIST v1.1
Progression-Free Survival (PFS) | Up to approximately 3 years
  Progression-free survival per RECIST v1.1
Number of patients with AEs in Phase 2 | Up to approximately 3 years
  Incidence and severity of treatment-emergent AEs and serious AEs as assessed by CTCAE v5
Changes in vital signs in Phase 2 | Up to approximately 3 years
  Number of patients with clinically significant changes in vital signs
Changes in clinical laboratory values in Phase 2 | Up to approximately 3 years
  Number of patients with clinically significant changes in clinical laboratory test values
Overall Survival (OS) in Phase 2 | Up to approximately 3 years
  OS is defined as time from enrollment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc., Study Director — Revolution Medicines, Inc.
Locations (53):
- United States (21):
  - City of Hope, Duarte, California
  - UC IRVINE Health, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Columbia University, New York, New York
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institue, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson, Houston, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT Oncology San Antonio, San Antonio, Texas
  - START Texas, San Antonio, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
- France (8):
  - West Cancer Institute, Angers
  - Institut Bergonie, Bordeaux
  - Hospital Louise Pradel, Bron
  - Oscar Lambret Center of Lillle, Lille
  - Centre Leon Berard, Lyon
  - Cancer Institute of Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Institute of Cancer of Strasbourg, Strasbourg
- Germany (4):
  - Universitäts Klinikum Köln, Cologne
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Krankenhaus Bethanien Moers, Moers
  - Klinkum Nurnberg Paracelsus Medical Unviersity, Nuremberg
- Italy (7):
  - Department of Medical Oncology - Azienda Ospedaliero Uniersitaria delle Marche, Ancona
  - Centro Di Riferimento Oncologico, Aviano
  - Institute Romagnolo per lo Studio Tumori, Meldola
  - Niguarda Cancer Center, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione "G. Pascale", Napoli
  - San Luigi Hospital, Orbassano
  - AUSL Romagna - S.M. delle Croci Hospital, Ravenna
- Netherlands Cancer Institute Antoni van Leeuwenhoek, Amsterdam, Netherlands
- Pan American Center for Oncology Trials, San Juan, Puerto Rico
- Spain (11):
  - START Barcelona - Hospital HM Nou Delfos, Barcelona
  - Institut Catala d'Oncologia Hospital, Barcelona
  - University Clinic of Navarra, Madrid
  - Fundacion MD Anderson Cancer Center, Madrid
  - START Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - NEXT Oncology - Quirónsalud Madrid University Hospital, Madrid
  - University Clinic of Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - La Fe University and Polytechnic Hospital, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cregg J, Edwards AV, Chang S, Lee BJ, Knox JE, Tomlinson ACA, Marquez A, Liu Y, Freilich R, Aay N, Wang Y, Jiang L, Jiang J, Wang Z, Flagella M, Wildes D, Smith JAM, Singh M, Wang Z, Gill AL, Koltun ES. Discovery of Daraxonrasib (RMC-6236), a Potent and Orally Bioavailable RAS(ON) Multi-selective, Noncovalent Tri-complex Inhibitor for the Treatment of Patients with Multiple RAS-Addicted Cancers. J Med Chem. 2025 Mar 27;68(6):6064-6083. doi: 10.1021/acs.jmedchem.4c02314. Epub 2025 Mar 8. PMID 40056080